CLINICAL TRIAL: NCT03771001
Title: 5Minutes4Myself: A Wellness Program for Caregivers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding to rebuild the app
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-1004
Record Dates: First submitted 2018-11-30; First posted 2018-12-10 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Autism; Stress; Autism Spectrum Disorder
Keywords: Wellness; Caregivers; Lifestyle; Stressor
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Convenience sample participants (Other): In this feasibility study all participants will receive the intervention.
  Interventions: Other: Motivational Interviewing coaching and habit-building app

INTERVENTIONS:
Other: Motivational Interviewing coaching and habit-building app — Coaches will use a manualized motivational interviewing approach and participants' wellness promoting changes will be supported via a habit building app that also delivers a micro-mindfulness program

SUMMARY:
This research study refines a wellness program designed for caregivers of autistic children called 5Minutes4Myself and further investigates its feasibility. Participants will attend a workshop to consent, participate in focus groups on lifestyle issues, and complete a baseline survey. Participants will have an individualized consultation with a coach to develop their tailored wellness program and be introduced to an app that support habits to build wellness activities into their daily life. The app provides the participant with their goal profile, tailored reminders, weekly check-ins, and delivers a micro-mindfulness program. Coaches will check-in monthly with participants and work together to modify their program as desired. After 4-6 months, participants will gather for a closing workshop to discuss their lifestyle and to evaluate the program. Pre-/post-surveys will examine health, well-being, stress, depression, and mindfulness. The app usability will be assessed using the Modified Systems Usability Scale (MSUS) as well as usage data.

DETAILED DESCRIPTION:
This study is designed to:

1. Conduct focus groups with caregivers of autistic children to understand specific stressors that they experience;
2. Gather baseline data including surveys of health and well-being;
3. Administer an individualized wellness program by using motivational interviews (MI) to individually tailor the program for each participant, train participants to use an app designed to support the adoption of lifestyle changes;
4. Coach participants over the 4-6 months of their program; and
5. Assess the usability of the app and the impact of the wellness program on caregiver's health and well-being.

Participants will be invited to the University of Wisconsin-Madison campus or participate online where they will:

1. complete baseline surveys of physical and mental health, mindfulness, stress, and wellbeing (Center for Epidemiology Depression Scale -Revised; Five Facet Mindfulness Questionnaire; Perceived Stress Scale; Psychological Well-being Scale; Rand Short Form-36),
2. get introduced to the study procedures and research team (Principal Investigator, Researcher, and MI-trained Masters-level occupational therapy and counseling graduate students); and
3. participate in focus groups to introduce the 5Minutes4Myself program, offer data on current lifestyles, and receive training on how to use the app

Participants will be assigned coaches. They will work together in an initial lifestyle coaching session and continue meeting monthly for 4-6 months. To assess the fidelity of the coaching sessions, motivation interviewing sessions (initial and monthly) will be audio-- or video--taped to assess fidelity via the Motivational Interviewing Treatment Integrity tool (MITI). Participants will be asked to complete an assessment of their satisfaction with the coaching. Data will be archived for the ongoing project.

The coaches will use Motivational Interviewing strategies to identify barriers to implementing the mindfulness program, foster commitment talk, and elicit the participant's strategy for implementing the mindfulness program in their daily life. Participants may request additional consultation through the weekly app goal check-in or via email.

The app will host all baseline surveys allowing them to be completed electronically. The baseline surveys will be completed prior to the first coaching session. The app will also be used as a "habit builder" providing personalized notifications as to when a goal activity will be created, will have goal check ins for each goal, and will collect usage data for audio mindfulness podcasts that are part of the program. Usage data will show how often and for how long participants listened to a podcast during the intervention.

After completing the 4-6 month intervention, participants will return for another workshop that will include:

1. Completion of Focus Group;
2. Re-administration of 'baseline' surveys (now considered 'post-intervention');
3. Assessing the usability of the app via the MSUS; and

ELIGIBILITY:
Inclusion Criteria:

1. Primary caregivers for child with autism OR primary caregiver of grandchild
2. Child cared for is between 8 - 21 for caregivers of children with autism and 5-21 years of age for grandchildren being parented by grandparents
3. Willingness to commit sufficient time to participate in the program
4. Desire to participate in a lifestyle/wellness program

Exclusion Criteria:

1. Caregivers of children younger than 8 years of age or older than 21 years of age for sample of parents of children with autism and Caregiver of child younger than 5 or older than 21 for grandparents parenting grandchildren
2. Caregivers with significant mental illness (except for those diagnosed or treated for depression who will be included)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
SF-36 Questionnaire | Up to 6 months
  Survey assessing mental and physical health
Perceived Stress Scale | Up to 6 months
  The Perceived Stress Scale is a measure of the degree to which the participant perceives their life as stressful. A series of 10 questions are asked to which the participant answers either: 0 = Never; 1 = Almost Never; 2 = Sometimes; 3 = Fairly Often; 4 = Very Often. The scoring for positively worded questions is calculated by reversing the response (0=4, 1=3, 2=2, 3=1, 4=0). Higher total scores indicate more perceived stress.
Ryff's Psychological Well-Being Scale | Up to 6 months
  Ryff's Psychological Well-Being is a self-reported scale to assess well-being. Participants respond to various statements about autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance and indicate how true each statement is of them on a 6-point Likert scale. Higher scores are representative of greater sense of well-being.
Center for Epidemiological Depression Scale-Revised | Up to 6 months
  The Center for Epidemiological Depression Scale (Revised; CESD-R) is a self-reported assessment where the participant answers 20 questions about how they have felt or behaved over the past 1-2 weeks. It is scored: 0 = Not at All or less than 1 day; 1 = 1-2 days; 2 = 3-4 days; 3 = 5-7 days; 4 = nearly every 5 for 2 weeks. Higher scores indicate greater depressive state.
Five facets of Mindfulness Questionnaire | Up to 6 months
  Assess degree of mindfulness
Modified System Usability Scale | Up to 6 months
  The Modified System Usability Scale is a 10 item questionnaire where the participants have 5 responses ranging from Strongly Agree to Strongly Disagree. The responses are assigned values such that the total score ranges from 1-100 with higher scores indicating increased usability.
Participant Feedback | Up to 6 months
  An important outcome measure will be direct participant feedback. Program feedback will be collected via focus group participation.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Larson, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Community Sites, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No